CLINICAL TRIAL: NCT03947359
Title: Effect of Thoracic Diameter and Food Intake on Fibroscan® Results: Comparison of the S - and M-probes
Brief Title: Effect of Thoracic Diameter and Food Intake on Fibroscan® Results
Acronym: FS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Fibroscan_V1
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Liver Stiffness

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with a thoracic diameter < 75 cm (Other): Measurement of liver stiffness before and after a standardized meal with different probes
  Interventions: Diagnostic Test: Fibroscan Touch 502 M probe; Diagnostic Test: Fibroscan Touch 502 S probe
- Participants with a thoracic diameter >75 cm (Other): Measurement of liver stiffness before and after a standardized meal with different probes
  Interventions: Diagnostic Test: Fibroscan Touch 502 M probe; Diagnostic Test: Fibroscan Touch 502 S probe

INTERVENTIONS:
Diagnostic Test: Fibroscan Touch 502 M probe — Measurement of liver stiffness
Diagnostic Test: Fibroscan Touch 502 S probe — Measurement of liver stiffness

SUMMARY:
The study aims to deliver scientific data regarding the accuracy of the two different-sized Fibroscan® probes on patients with different thoracic diameter to gain more knowledge of the handling and measuring quality of the Fibroscan® as a diagnostic device and also to see if one probe is enough to measure a wider spectrum of patients leading to cost reduction for equipment such as additional probes.

Furthermore the study aims to analyze the effect of food intake on liver-stiffness measurements with the S-probe on children to shorten fasting periods. It is hypothesized that the fasting periods before a Fibroscan® measurement may be shortened, which is of special importance in smaller children.

DETAILED DESCRIPTION:
The Fibroscan® (Echosens, France) is an ultrasound-based, non-invasive and non-painful diagnostic device which also has no complications and can be repeated easily to measure liver-stiffness by transient elastography. The company's device was first released and put on the market in 2003. The device can measure liver stiffness and liver fat content (controlled attenuation parameter CAP).

It is used for the identification and graduation of liver pathologies such as fibrosis and cirrhosis and it can be used on adults and children alike. Therefore patients with chronic liver diseases such as hepatitis C, hepatitis B, alcoholic liver disease as well as metabolic steatohepatitis and different biliary diseases can be examined with it.

Currently the standard procedure for grading fibrosis and cirrhosis still is the liver biopsy, however studies have compared the two procedures in context with different liver conditions like non-alcoholic fatty liver disease or hepatitis C and partially demonstrated that in terms of measuring liver-stiffness the Fibroscan® can rival the liver biopsy.

Usually the Fibroscan® measurements are performed using different probes that vary in frequency and penetration depth depending on the thoracic diameter of the patient. These probes are then applied in an intercostal space on the right side on the level of the liver.

The company Echosens that is producing the currently used model of the Fibroscan® alongside its different-sized probes claims that their S-sized probe is to be used for patients with a thoracic diameter below 75 cm and that their M-sized probe for patients above 75 cm diameter because otherwise the results would not be accurate. The company claims that using the M-sized probe on a patient with a thoracic diameter below 75 cm would cause wrong measurements. However, there is no data or studies that actually have compared the S- and the M- probe to each other and therefore the accuracy of the statement from Echosens is scientifically yet to be confirmed. So far only data on comparison of the M and XL-probe have been published.

Furthermore, food intake seems to impact on Fibroscan® -measurements. It has been already proven in past studies that food intake indeed has an effect on liver-stiffness and therefore influences the quality of Fibroscan® -measurements. All these studies revealed that it is the best to measure the patients while in a fasting condition for several hours. However, these studies all were performed on adults with different kinds of liver-diseases using the M-probe. So far, no data on the impact of food intake on measurements with the S-probe have been published.

Since it is to be expected that because of its attributes transient elastography will gain even more importance as a diagnostic device in the future, it is very significant to produce as much of valid data as possible.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 for the adult Population

Age 11-18 for the paediatric population

Informed consent

No history of liver disease

Thoracic diameter >45 cm

Exclusion Criteria:

Acute or chronic liver disease

Any other disease or circumstance that may impact on the result of the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Liver stiffness | baseline
  Comparison of liver stiffness measurements at baseline with M- and S- probe

SECONDARY OUTCOMES:
Liver stiffness | 120 minutes
  Measurement of liver stiffness measurements with M- probe after a standardized meal
Liver stiffness | 120 minutes
  Measurement of liver stiffness measurements with S- probe after a standardized meal
Liver fat content | baseline
  Controlled attenuation parameter measured with M probe
Liver fat content | 120 minutes
  Controlled attenuation parameter measured with S probe

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No